CLINICAL TRIAL: NCT02169388
Title: Effects of Gut Microflora on the Immune and Nutritional Status of CRC Patients After Chemotherapy
Brief Title: Intestinal Microflora in Colorectal Cancer (CRC) After Chemotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2014SDU-QILU-G03
Record Dates: First submitted 2014-06-04; First posted 2014-06-23 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Gastrointestinal Neoplasms; Colorectal Cancer; Effects of Chemotherapy; Tumor Immunity; Malnutrition
Keywords: Gut microflora; colorectal cancer; Chemotherapy; Immunity; Nutrition
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Malnutrition | interventions — Probiotics; phosphatidyltransferase, Clostridium butyricum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): Microbial composition using Probiotic，3 capsules / times, 2 times / day for 4 weeks
  Interventions: Drug: Probiotic
- placebo (Placebo Comparator): Microbiota modulation using placebo，3 capsules / times, 2 times / day for 4 weeks
  Interventions: Drug: placebo（for probiotic）

INTERVENTIONS:
Drug: Probiotic — Microbial composition using probiotic
  Other Names: containing; （ clostridium butyricum）
  Arms: Probiotic
Drug: placebo（for probiotic） — microbiota modulation using placebo
  Arms: placebo

SUMMARY:
Probiotics modulate the gut microflora and immune status in CRC,which can reduce the side effects of chemotherapy such as diarrhea,infection,neutropenia etc.

DETAILED DESCRIPTION:
Chemotherapy destroys the intestinal mucosal barrier, affects intestinal flora, causing bacterial translocation, infection and other complications; Probiotics may restore the intestinal immunity, mucosal barrier, and nutrient absorption.The adverse effects of chemotherapy and the malnutrition status may be relieved via probiotic administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for chemotherapy after radical resection of colorectal cancer

Exclusion Criteria:

* Palliative resection of colorectal cancer
* Antibiotic,probiotic or prebiotic usage within 1months
* Other malignancy
* History of other abdominal surgery
* Coagulopathy or bleeding disorders
* Pregnant or breast-feeding(for females)
* Impaired liver or renal function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-10 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Composition of Microorganisms in stool after probiotic intervention | 5 months
  Primary coordination of fecal samples' 16s rDNA (ribosomal DNA) will be compared between two Groups using Braycurtis distance based Primary coordination analysis (PCoA).
Short-chain fatty acids in feces of patients after chemotherapy | 5 months
  The total concentration of Short-chain fatty acids in the in feces of patients after chemotherapy.
Frequency and severity of Adverse effects during Chemotherapy | 5 months
  Adverse effects includes vomiting, nausea, diarrhea and abdominal pain.

SECONDARY OUTCOMES:
The observed changes in immune status after chemotherapy | 5 month
  Immune status indexes include percentage of Neutrophils, total lymphocytes, lymphocyte subgroups, plasma immunoglobulin level, CRP (C reactive protein).
The observed changes in nutritional status after chemotherapy | 5 months
  Nutritional status indexes include BMI, percentage of body weight changes, plasma albumin and prealbumin.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD.PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China